CLINICAL TRIAL: NCT02531100
Title: PolyPid, Ltd. Pilot Study of the BonyPid-500TM Bone Graft Substitute
Brief Title: BonyPid-500TM Bone Graft Substitute Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PolyPid Ltd. (Industry)
Collaborators: MIS Implant Technologies, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BonyPid-201
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Peri Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BonyPid-500TM implantation (Experimental): Standard of care (SOC) treatment (Manual and ultrasonic debridement and surface decontamination) followed by BonyPid-500TM implantation.
  Interventions: Device: BonyPid 500TM implantation concomitantly to SOC treatment; Other: SOC treatment only
- SOC treatment (Other): Standard of care treatment (Manual and ultrasonic debridement and surface decontamination) only
  Interventions: Other: SOC treatment only

INTERVENTIONS:
Device: BonyPid 500TM implantation concomitantly to SOC treatment — BonyPid 500TM implantation concomitantly to SOC treatment
  Arms: BonyPid-500TM implantation
Other: SOC treatment only — Standard of care treatment (Manual and ultrasonic debridement, and surface decontamination)

SUMMARY:
This study is designed to assess the safety and effectiveness of BonyPid-500TM implantation for intrabony peri-implantitis defects.

BonyPid-500™ is a bone graft substitute, which contains an antibiotic drug - doxycycline, and is intended for filling and reconstruction of bone defects caused by peri-implantitis.

DETAILED DESCRIPTION:
This is a pilot, randomized, single-blind, two arm controlled, multicenter study in subjects undergoing surgical treatment for peri-implantitis disease. Eligible subjects will undergo a surgical treatment and be randomly assigned during surgical intervention (after flap opening) in a 1:1 ratio to adjunct BonyPid-500TM implantation or no BonyPid-500TM implantation.

Randomization will be stratified by site and number of eligible implants, i.e., single or multiple.

The study population includes male and female subjects, 20 - 80 years of age at screening, diagnosed with peri-implantitis and recommended for surgical treatment of peri-implantitis disease.

Up to 77 subjects will be enrolled to this study which will be conducted in two medical centers in Israel.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects, 20 - 80 years of age at screening.
* Females of childbearing potential must have a negative urine pregnancy test before radiographs, dental hygienist cleaning, and surgical procedure (Note: Females of childbearing age must agree to use a highly effective method of contraception consistently and correctly for the duration of the study period).
* Subjects with a minimum of one osseo-integrated implant with peri-implantitis.
* Subjects with at least one eligible implant within the surgical area.
* Subjects with bleeding on probing of selected implant with or without suppuration.
* Subjects with selected implant(s) having radiographic evidence, according to X-rays, of:

  1. Intrabony defect
  2. Bone loss ≥ 3 mm
  3. Minimum of 2 mm of bone at implant apex.
* Subjects must be willing and able to provide a written informed consent prior to any protocol specific procedures being performed and comply with protocol requirements.

Exclusion Criteria:

* Subjects with hydroxyapatite (HA) coated implants, titanium plasma spray implants.
* Subjects with a distance between implants < 3 mm, or < 2 mm between implant and tooth.
* Subjects with implants supporting removable dentures.
* Subjects presenting with severe active periodontitis.
* Subjects with poor oral hygiene.
* Subjects with selected implant(s) with radiographic evidence of horizontal bone loss only.
* Subjects suffering from Type 1 (insulin dependent) diabetes; or uncontrolled Type 2 diabetes. Diabetic subjects must provide a statement from a physician regarding the status of diabetes, in addition to a recent (within 3 months) documented Hemoglobin (Hgb) A1c blood test of < 6.5%.
* Pregnant women or women who intend to become pregnant during the study period, or breastfeeding women.
* Subjects with known allergy or contraindication to tetracycline(s).
* Subjects who are current smokers or who were smokers within 3 months prior to screening.
* Subjects who were under oral or local antibiotic therapy in the last 4 weeks prior to study enrollment.
* Subjects treated for at least 2 weeks with any medication known to affect soft tissue condition within one month prior to study enrollment (e.g., Phenytoin, Cyclosporine, Coumadin, and NSAIDs).
* Subjects treated with Oral or IV use of doxycycline in the last four weeks prior to screening.
* Subjects with presence of active systemic infectious diseases such as: hepatitis, HIV, or a history of tuberculosis.
* Subjects with any condition, which in the opinion of the Investigator, would place the subject at risk or influence the conduct of the study or interpretation of results.
* Subjects who are incapable of following the study schedule for any reason, per the Investigator's discretion.
* Subjects who are currently enrolled, recently participated (within 30 days prior to screening), or planning to enroll in another study that may conflict with protocol requirements or may confound the subject results in this trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Safety: AEs (adverse events) as reported by the subject or observed by the Investigator, | 12 months
  All AEs including any change in medical or dental status.
Effectiveness: the change in Pocket Probing Depth (cPPD) from baseline to 6 months, measured in mm. | 6 months
  The primary effectiveness endpoint of the study is the change in Pocket Probing Depth (cPPD) from baseline to 6 months, measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Belotserkovsky, Study Director — Sponsor GmbH
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: No